CLINICAL TRIAL: NCT00899470
Title: Bioequivalence Study of the Fixed Dose Combination of 2.5 mg Saxagliptin and 500 mg Metformin Immediate Release (IR) Tablet Relative to 2.5 mg Saxagliptin Tablet and 500 mg Metformin IR Tablet Co-administered to Healthy Subjects in a Fasted and in a Fed State
Brief Title: Bioequivalence Study of Saxagliptin and Glucophage Combination Formulations in Healthy Subjects (A)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CV181-081
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2011-03-25 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- S+ M, (fasted)> S/M (fed)> S/M (fasted)>S+M (fed) (Experimental): Participants were randomized to receive oral co-administration of a 2.5 mg tablet of saxagliptin plus a 500 mg tablet of metformin immediate release (IR) under fasted conditions (S + M [fasted]) followed by a fixed dose combination (FDC) tablet of 2.5 mg saxagliptin/500 mg metformin IR under fed conditions (S/M [fed]) followed by S/M under fasting conditions (S/M [fasted]) followed by S + M under fed conditions (S + M [fed])
  Interventions: Drug: Co-administration of Saxagliptin and Metformin IR, Fasted; Drug: Saxagliptin/Metformin, Fasting; Drug: Co-administration of Saxagliptin and Metformin IR, Fed; Drug: Saxagliptin/Metformin, Fed
- S/M (fasted)> S+M (fasted)> S+M (fed)> S/M (fed) (Experimental): Participants were randomized to receive S/M (fasted) followed by S + M (fasted) followed by S + M (fed) followed by S/M (fed)
  Interventions: Drug: Co-administration of Saxagliptin and Metformin IR, Fasted; Drug: Saxagliptin/Metformin, Fasting; Drug: Co-administration of Saxagliptin and Metformin IR, Fed; Drug: Saxagliptin/Metformin, Fed
- S+M (fed)> S/M (fasted) >S/M (fed)> S+M (fasted) (Experimental): Participants were randomized to receive S + M (fed) followed by S/M (fasted) followed by S/M (fed) followed by S+M (fasted)
  Interventions: Drug: Co-administration of Saxagliptin and Metformin IR, Fasted; Drug: Saxagliptin/Metformin, Fasting; Drug: Co-administration of Saxagliptin and Metformin IR, Fed; Drug: Saxagliptin/Metformin, Fed
- S/M (fed)> S+M (fed)> S+M (fasted)> S/M (fasted) (Experimental): Participants were randomized to receive S/M (fed) followed by S+M (fed) followed by S+M (fasted) followed by S/M (fasted)
  Interventions: Drug: Co-administration of Saxagliptin and Metformin IR, Fasted; Drug: Saxagliptin/Metformin, Fasting; Drug: Co-administration of Saxagliptin and Metformin IR, Fed; Drug: Saxagliptin/Metformin, Fed

INTERVENTIONS:
Drug: Co-administration of Saxagliptin and Metformin IR, Fasted — Participants received oral co-administration of a 2.5 mg tablet of saxagliptin and a 500 mg tablet of metformin immediate release (IR) under fasted conditions
  Other Names: Onglyza
Drug: Saxagliptin/Metformin, Fasting — Participants received a single oral dose of a fixed dose combination (FDC) tablet of 2.5 mg saxagliptin/500 mg metformin IR under fasting conditions
  Other Names: Onglyza; Glucophage
Drug: Co-administration of Saxagliptin and Metformin IR, Fed — Participants received oral co-administration of a 2.5 mg tablet of saxagliptin and a 500 mg tablet of metformin immediate release (IR) under fed conditions
Drug: Saxagliptin/Metformin, Fed — Participants received a single oral dose of a fixed dose combination (FDC) tablet of 2.5 mg saxagliptin/500 mg metformin IR under fed conditions

SUMMARY:
To demonstrate bioequivalence of a 2.5 mg saxagliptin/500 mg metformin (glucophage) immediate release (IR) fixed dose combination (FDC) tablet to the 2.5 mg saxagliptin tablet and 500 mg metformin IR tablet co-administered to healthy subjects in a fasted and in a fed state.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 19 to 45 inclusive
* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 32 kg/m2, inclusive. BMI = weight (kg)/ [height (m)]2

Exclusion Criteria:

* Women of child-bearing potential (WOCBP) who are unwilling or unable to use acceptable barrier methods (condoms and spermicides) to avoid pregnancy for the entire study period and for up to 8 weeks after the last dose of investigational product
* Any significant acute or chronic medical illness
* Current or recent (within 3 months) gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* History of allergy to Dipeptidyl peptidase 4 (DPP4) inhibitor or related compounds
* History of allergy or intolerance to metformin or other similar acting agents
* Prior exposure to saxagliptin
* Prior exposure to metformin within 3 months of study drug administration.
* Estimated creatinine clearance (Clcr) of < 80ml/min using the Cockcroft Gault formula

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Mds Pharma Services, Lincoln, Nebraska, United States

REFERENCES:
- [Derived] Upreti VV, Keung CF, Boulton DW, Chang M, Li L, Tang A, Hsiang BC, Quamina-Edghill D, Frevert EU, Lacreta FP. Bioequivalence of saxagliptin/metformin immediate release (IR) fixed-dose combination tablets and single-component saxagliptin and metformin IR tablets in healthy adult subjects. Clin Drug Investig. 2013 May;33(5):365-74. doi: 10.1007/s40261-013-0075-z. PMID 23549864
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 85 participants were enrolled and 24 were treated on study. 61 participants discontinued before randomization and treatment due to: no longer meeting study criteria (n=36), withdraw of consent (n=3), study was full (n=15), participant did not call for results (n=1), completed alternate status (n=5), or did not show for check-up (n=1)
Groups:
- S+M (Fasted)> S/M (Fed)> S/M (Fasted)>S+M (Fed): Participants were randomized to receive oral co-administration of a 2.5 mg tablet of saxagliptin plus a 500 mg tablet of metformin immediate release (IR) under fasted conditions (S + M [fasted]) followed by a fixed dose combination (FDC) tablet of 2.5 mg saxagliptin/500 mg metformin IR under fed conditions (S/M [fed]) followed by S/M under fasting conditions (S/M [fasted]) followed by S + M under fed conditions (S + M [fed])
Period: First Therapy
Arm/Group | S+M (Fasted)> S/M (Fed)> S/M (Fasted)>S+M (Fed) | S/M (Fasted)> S+M (Fasted)> S+M (Fed)> S/M (Fed) | S+M (Fed)> S/M (Fasted) >S/M (Fed)> S+M (Fasted) | S/M (Fed)> S+M (Fed)> S+M (Fasted)> S/M (Fasted)
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: First Washout Period
Arm/Group | S+M (Fasted)> S/M (Fed)> S/M (Fasted)>S+M (Fed) | S/M (Fasted)> S+M (Fasted)> S+M (Fed)> S/M (Fed) | S+M (Fed)> S/M (Fasted) >S/M (Fed)> S+M (Fasted) | S/M (Fed)> S+M (Fed)> S+M (Fasted)> S/M (Fasted)
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Second Therapy
Arm/Group | S+M (Fasted)> S/M (Fed)> S/M (Fasted)>S+M (Fed) | S/M (Fasted)> S+M (Fasted)> S+M (Fed)> S/M (Fed) | S+M (Fed)> S/M (Fasted) >S/M (Fed)> S+M (Fasted) | S/M (Fed)> S+M (Fed)> S+M (Fasted)> S/M (Fasted)
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Second Washout
Arm/Group | S+M (Fasted)> S/M (Fed)> S/M (Fasted)>S+M (Fed) | S/M (Fasted)> S+M (Fasted)> S+M (Fed)> S/M (Fed) | S+M (Fed)> S/M (Fasted) >S/M (Fed)> S+M (Fasted) | S/M (Fed)> S+M (Fed)> S+M (Fasted)> S/M (Fasted)
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Third Therapy
Arm/Group | S+M (Fasted)> S/M (Fed)> S/M (Fasted)>S+M (Fed) | S/M (Fasted)> S+M (Fasted)> S+M (Fed)> S/M (Fed) | S+M (Fed)> S/M (Fasted) >S/M (Fed)> S+M (Fasted) | S/M (Fed)> S+M (Fed)> S+M (Fasted)> S/M (Fasted)
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Third Washout
Arm/Group | S+M (Fasted)> S/M (Fed)> S/M (Fasted)>S+M (Fed) | S/M (Fasted)> S+M (Fasted)> S+M (Fed)> S/M (Fed) | S+M (Fed)> S/M (Fasted) >S/M (Fed)> S+M (Fasted) | S/M (Fed)> S+M (Fed)> S+M (Fasted)> S/M (Fasted)
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Therapy
Arm/Group | S+M (Fasted)> S/M (Fed)> S/M (Fasted)>S+M (Fed) | S/M (Fasted)> S+M (Fasted)> S+M (Fed)> S/M (Fed) | S+M (Fed)> S/M (Fasted) >S/M (Fed)> S+M (Fasted) | S/M (Fed)> S+M (Fed)> S+M (Fasted)> S/M (Fasted)
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Treated Participants: Participants were randomized to received 1 of 4 treatments 1)oral co-administration of a 2.5 mg tablet of saxagliptin and a 500 mg tablet of metformin immediate release (IR) under fasted conditions, 2) a fixed dose combination (FDC) tablet of 2.5 mg saxagliptin/500 mg metformin IR under fasting conditions, 3) oral co-administration of a 2.5 mg tablet of saxagliptin and a 500 mg tablet of metformin immediate release (IR) under fed conditions, or 4) a fixed dose combination (FDC) tablet of 2.5 mg saxagliptin/500 mg metformin IR under fed conditions. Participants received all 4 treatments in 1 of 4 sequences: 1-4-2-3, 2-1-3-4, 3-2-4-1, or 4-3-1-2, with a washout period between treatments of at least 1 week.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Saxagliptin Mean Maximum Observed Plasma Concentration (Cmax)
Description: Cmax of single-dose saxagliptin (2.5 mg), either coadministered with metformin IR (500 mg), or administered as FDC 2.5 mg saxagliptin/500 mg metformin IR, under fasted and fed conditions.
Time Frame: Day 1: 0 hr, 0.25 hr, 0.5 hr, 0.75 hr, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, 12 hr, 18 hr, Day 2: 0 hr, 12 hr, Day 3: 0 hr
Population: PK data set, all participants who received study drug
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Coadministration of Saxagliptin and Metformin IR (Fasted): Participants received oral coadministration of a 2.5 mg tablet of saxagliptin and a 500 mg tablet of metformin immediate release (IR) under fasted conditions
- Saxagliptin/Metformin FDC (Fasted): Participants received a single oral dose of a fixed-dose combination (FDC) tablet of 2.5 mg saxagliptin/500 mg metformin IR under fasting conditions
- Coadministration of Saxagliptin and Metformin IR (Fed): Participants received oral coadministration of a 2.5 mg tablet of saxagliptin and a 500 mg tablet of metformin IR under fed conditions
- Saxagliptin/Metformin FDC (Fed): Participants received a single oral dose of an FDC tablet of 2.5 mg saxagliptin/500 mg metformin IR under fed conditions
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/mL | 8.57 (2.572) | 8.61 (2.266) | 11.36 (2.875) | 11.51 (3.781)
Statistical Analysis 1: Comparison: Coadministration of Saxagliptin and Metformin IR (Fasted) vs Saxagliptin/Metformin FDC (Fasted); To demonstrate bioequivalence (BE) of FDC tablets (Test) versus co-administration of saxagliptin and metformin IR tablets (Reference) formulations in fasted state, linear mixed model analysis was performed on log(Cmax) of saxagliptin. Factors in the model were sequence, period and treatment as fixed effects, and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — If no difference between bioavailabilities of saxagliptin from FDC tablet vs. co-administration of saxagliptin tablet and metformin (fasted condition), then 20 subjects provided 97% power to conclude BE with respect to Cmax of saxagliptin. If 5% difference then 20 subjects provided 93% power to conclude BE with respect to Cmax of saxagliptin; Mixed Models Analysis; Bioequivalence=90% confidence intervals (CIs) for the test; Geometric Mean Ratio, Test vs. Reference = 1.011, 90% CI 2-sided [0.940 to 1.088] — For Cmax of saxagliptin, the point estimate and 90% CI were calculated for the ratio of the geometric mean of the Test formulation in fasted state: the geometric mean of the Reference formulation in fasted state
Statistical Analysis 2: Comparison: Coadministration of Saxagliptin and Metformin IR (Fed) vs Saxagliptin/Metformin FDC (Fed); To demonstrate BE of FDC tablets (Test) versus co-administration of saxagliptin and metformin IR tablets (Reference) formulations in fed state, linear mixed model analysis was performed on log(Cmax) of saxagliptin. Factors in the model were sequence, period and treatment as fixed effects, and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — If no difference between bioavailabilities of saxagliptin from FDC tablet vs. co-administration of saxagliptin tablet and metformin (fed condition), then 20 subjects provided 97% power to conclude BE with respect to Cmax of saxagliptin. If 5% difference then 20 subjects provided 93% power to conclude BE with respect to Cmax of saxagliptin; Bioequivalence=90% CIs for the test; Geometric Mean Ratio, Test vs Reference = 0.999, 90% CI 2-sided [0.929 to 1.075] — For Cmax of saxagliptin, the point estimate and 90% CI were calculated for the ratio of the geometric mean of the Test formulation in fed state: the geometric mean of the Reference formulation in fed state

2. Primary Outcome: Saxagliptin Mean Area Under the Plasma Concentration Time Curve From Time Zero To Time of Last Quantifiable Concentration (AUC [0-T]}
Description: AUC (0-T) for single-dose saxagliptin (2.5 mg), either coadministered with metformin IR (500 mg), or administered as FDC 2.5 mg saxagliptin/500 mg metformin IR, under fasted and fed conditions.
Time Frame: as for outcome 1
Population: PK data set, all participants who received study drug
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng*h/mL | 48.57 (12.864) | 49.69 (12.330) | 54.59 (12.407) | 55.83 (12.735)
Statistical Analysis 1: Comparison: Coadministration of Saxagliptin and Metformin IR (Fasted) vs Saxagliptin/Metformin FDC (Fasted); To demonstrate BE of FDC tablets (Test) versus co-administration of saxagliptin and metformin IR tablets (Reference) formulations in fasted and fed states, linear mixed model analysis was performed on log[AUC(0-T)] of saxagliptin. Factors in the model were sequence, period and treatment as fixed effects, and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — If no difference between bioavailabilities of saxagliptin from FDC tablet vs. co-administration of saxagliptin tablet and metformin (fasted condition), then 20 subjects provided 99% power to conclude BE with respect to AUC(INF) of saxagliptin. If 5% difference then 20 subjects provided 99% power to conclude BE with respect to AUC(INF) of saxagliptin; Mixed Models Analysis; Bioequivalence=90% CIs for the test; Geometric Mean Ratio, Test vs. Reference = 1.029, 90% CI 2-sided [0.993 to 1.066] — For AUC(0-T) of saxagliptin, the point estimate and 90% CI were calculated for the ratio of the geometric mean of the Test formulation in fasted state: geometric mean of the Reference formulation in fasted state
Statistical Analysis 2: Comparison: Coadministration of Saxagliptin and Metformin IR (Fed) vs Saxagliptin/Metformin FDC (Fed); To demonstrate BE of FDC tablets (Test) versus co-administration of saxagliptin and metformin IR tablets (Reference) formulations in fed state, linear mixed model analysis was performed on log[AUC(0-T)] of saxagliptin. Factors in the model were sequence, period and treatment as fixed effects, and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — If no difference between bioavailabilities of saxagliptin from FDC tablet vs. co-administration of saxagliptin tablet and metformin (fed condition), then 20 subjects provided 99% power to conclude BE with respect to AUC(INF) of saxagliptin. If 5% difference then 20 subjects provided 99% power to conclude BE with respect to AUC(INF) of saxagliptin; Mixed Models Analysis; Bioequivalence=90% CIs for the test; Geometric Means Ratio = 1.021, 90% CI 2-sided [0.986 to 1.058] — For AUC(0-T) of saxagliptin, the point estimate and 90% CI were calculated for the ratio of the geometric mean of the Test formulation in fed state: the geometric mean of the Reference formulation in fed state

3. Primary Outcome: Saxagliptin Mean Area Under the Plasma Concentration Time Curve From Time Zero To Infinity (AUC [0-INF])
Description: as for outcome 2
Time Frame: as for outcome 1
Population: PK data set, all participants who received study drug
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng*h/mL | 50.66 (13.322) | 51.74 (12.736) | 56.56 (12.778) | 57.86 (13.222)
Statistical Analysis 1: Comparison: Coadministration of Saxagliptin and Metformin IR (Fasted) vs Saxagliptin/Metformin FDC (Fasted); To demonstrate BE of FDC tablets (Test) versus co-administration of saxagliptin and metformin IR tablets (Reference) formulations in fasted state, linear mixed model analysis was performed on log[AUC(INF)] of saxagliptin. Factors in the model were sequence, period and treatment as fixed effects, and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mixed Models Analysis; Bioequivalence=90% CIs for the test; Geometric Mean Ratio, Test vs. Reference = 1.027, 90% CI 2-sided [0.990 to 1.066] — For AUC(INF) of saxagliptin, the point estimate and 90% CI were calculated for the ratio of the geometric mean of the Test formulation in fasted state: geometric mean of the Reference formulation in fasted state
Statistical Analysis 2: Comparison: Coadministration of Saxagliptin and Metformin IR (Fed) vs Saxagliptin/Metformin FDC (Fed); To demonstrate BE of FDC tablets (Test) versus co-administration of saxagliptin and metformin IR tablets (Reference) formulations in fed state, linear mixed model analysis was performed on log[AUC(INF)] of saxagliptin and metformin. Factors in the model were sequence, period and treatment as fixed effects, and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; Mixed Models Analysis; Bioequivalence=90% CIs for the test; Geometric Means Ratio Test vs. Reference = 1.022, 95% CI 2-sided [0.985 to 1.060] — For AUC(INF) of saxagliptin, the point estimate and 90% CI were calculated for the ratio of the geometric mean of the Test formulation in fed state: the geometric mean of the Reference formulation in fed state

4. Primary Outcome: Saxagliptin Mean Plasma Half-life (T-half) and Mean Time of Maximum Observed Plasma Concentration (T-max)
Description: T-half and T-max for single-dose saxagliptin (2.5 mg), either coadministered with metformin IR (500 mg) or administered as FDC 2.5 mg saxagliptin/500 mg metformin IR, under fasted and fed conditions.
Time Frame: as for outcome 1
Population: PK data set, all participants who received study drug
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
hours
  T-half | 5.86 (1.367) | 5.55 (1.135) | 5.75 (1.119) | 5.72 (1.146)
  T-max | 1.78 (1.210) | 1.23 (0.829) | 1.37 (0.842) | 1.42 (0.862)

5. Primary Outcome: Metformin Mean Cmax
Description: Cmax of single-dose metformin IR (500 mg), either coadministered with saxagliptin (2.5 mg) or administerd as FDC 2.5 mg saxagliptin/500 mg metformin IR, under fasted and fed conditions.
Time Frame: as for outcome 1
Population: PK data set, all participants who received study drug
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/mL | 1030.22 (293.970) | 1042.52 (314.365) | 993.32 (198.653) | 1027.70 (208.974)
Statistical Analysis 1: Comparison: Coadministration of Saxagliptin and Metformin IR (Fasted) vs Saxagliptin/Metformin FDC (Fasted); To demonstrate BE of FDC tablets (Test) versus co-administration of saxagliptin and metformin IR tablets (Reference) formulations in fasted state, linear mixed model analysis was performed on log(Cmax) of metformin. Factors in the model were sequence, period and treatment as fixed effects, and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — If no difference between bioavailabilities of metformin from FDC tablet vs. co-administration of saxagliptin tablet and metformin (fasted and fed), then 20 subjects provided 98% power to conclude BE with respect to Cmax of metformin. If 5% difference then 20 subjects provided 93% power to conclude BE with respect to Cmax of metformin, respectively; Mixed Models Analysis; Bioequivalence=90% CIs for the test; Geometric Mean Ratio, Test vs. Reference = 1.009, 90% CI 2-sided [0.939 to 1.084] — For Cmax of metformin, the point estimate and 90% CI were calculated for the ratio of the geometric mean of the Test formulation in fasted state: geometric mean of the Reference formulation in fasted fed state
Statistical Analysis 2: Comparison: Coadministration of Saxagliptin and Metformin IR (Fed) vs Saxagliptin/Metformin FDC (Fed); To demonstrate BE of FDC tablets (Test) versus co-administration of saxagliptin and metformin IR tablets (Reference) formulations in fed state, linear mixed model analysis was performed on log(Cmax) of metformin. Factors in the model were sequence, period and treatment as fixed effects, and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — If no difference between bioavailabilities of metformin from FDC tablet vs. co-administration of saxagliptin tablet and metformin (fed), then 20 subjects provided 98% power to conclude BE with respect to Cmax of metformin. If 5% difference then 20 subjects provided 93% power to conclude BE with respect to Cmax of metformin; Mixed Models Analysis; Bioequivalence=90% CIs for the test; Geometric Mean Ratio, Test vs. Reference = 1.034, 90% CI 2-sided [0.962 to 1.111] — For Cmax of metformin, the point estimate and 90% CI were calculated for the ratio of the geometric mean of the Test formulation in fed state: the geometric mean of the Reference formulation in fed state

6. Primary Outcome: Metformin Mean AUC (0-T)
Description: AUC (0-T for single-dose metformin (500 mg), either coadministered with saxagliptin (2.5 mg) or administerd as FDC 2.5 mg saxagliptin/500 mg metformin IR, under fasted and fed conditions.
Time Frame: as for outcome 1
Population: PK data set, all participants who received study drug
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng*h/mL | 7403.01 (1822.749) | 7575.23 (1832.807) | 7176.78 (1216.854) | 7502.46 (1402.256)
Statistical Analysis 1: Comparison: Coadministration of Saxagliptin and Metformin IR (Fasted) vs Saxagliptin/Metformin FDC (Fasted); To demonstrate BE of FDC tablets (Test) versus co-administration of saxagliptin and metformin IR tablets (Reference) formulations in fasted state, linear mixed model analysis was performed on log[AUC(0-T)] of metformin. Factors in the model were sequence, period and treatment as fixed effects, and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — If no difference between bioavailabilities of metformin from FDC tablet vs. co-administration of saxagliptin tablet and metformin (fasted), then 20 subjects provided 99% power to conclude BE with respect to AUC(INF) of metformin. If 5% difference then 20 subjects provided 95% power to conclude BE with respect to AUC(INF) of metformin; Mixed Models Analysis; Bioequivalence=90% CIs for the test; Geometric Mean Ratio, Test vs. Reference = 1.024, 90% CI 2-sided [0.964 to 1.088] — For AUC(0-T) of metformin the point estimate and 90% CI were calculated for the ratio of the geometric mean of the Test formulation in fasted state: geometric mean of the Reference formulation in fasted state
Statistical Analysis 2: Comparison: Coadministration of Saxagliptin and Metformin IR (Fed) vs Saxagliptin/Metformin FDC (Fed); To demonstrate BE of FDC tablets (Test) versus co-administration of saxagliptin and metformin IR tablets (Reference) formulations in fed state, linear mixed model analysis was performed on log[AUC(0-T)] of metformin. Factors in the model were sequence, period and treatment as fixed effects, and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — If no difference between bioavailabilities of metformin from FDC tablet vs. co-administration of saxagliptin tablet and metformin (fed), then 20 subjects provided 99% power to conclude BE with respect to AUC(INF) of metformin. If 5% difference then 20 subjects provided 95% power to conclude BE with respect to AUC(INF) of metformin; Mixed Models Analysis; Bioequivalence=90% CIs for the test; Geometric Mean Ratio, Test vs. Reference = 1.042, 90% CI 2-sided [0.981 to 1.108] — For AUC(0-T) of metformin, the point estimate and 90% CI were calculated for the ratio of the geometric mean of the Test formulation in fed state: the geometric mean of the Reference formulation in fed state

7. Primary Outcome: Metformin Mean AUC(0-INF)
Description: AUC (0-INF) for single-dose metformin IR (500 mg), either coadministered with saxagliptin (2.5 mg) or administerd as FDC 2.5 mg saxagliptin/500 mg metformin IR, under fasted and fed conditions.
Time Frame: as for outcome 1
Population: PK data set, all participants who received study drug
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng*h/mL | 7494.67 (1792.921) | 7689.57 (1761.119) | 7246.89 (1215.675) | 7574.17 (1397.335)
Statistical Analysis 1: Comparison: Coadministration of Saxagliptin and Metformin IR (Fasted) vs Saxagliptin/Metformin FDC (Fasted); To demonstrate BE of FDC tablets (Test) versus co-administration of saxagliptin and metformin IR tablets (Reference) formulations in fasted state, linear mixed model analysis was performed on log[AUC(INF)] of metformin. Factors in the model were sequence, period and treatment as fixed effects, and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — If no difference between bioavailabilities of metformin from FDC tablet vs. co-administration of saxagliptin tablet and metformin (fasted ), then 20 subjects provided 99% power to conclude BE with respect to AUC(INF) of metformin. If 5% difference then 20 subjects provided 95% power to conclude BE with respect to AUC(INF) of metformin; Mixed Models Analysis; Bioequivalence=90% CIs for the test; Geometric Mean Ratio, Test vs. Reference = 1.029, 90% CI 2-sided [0.973 to 1.088] — For AUC(INF) of metformin, the point estimate and 90% CI were calculated for the ratio of the geometric mean of the Test formulation in fasted state: the geometric mean of the Reference formulation in fasted state
Statistical Analysis 2: Comparison: Coadministration of Saxagliptin and Metformin IR (Fed) vs Saxagliptin/Metformin FDC (Fed); To demonstrate BE of FDC tablets (Test) versus co-administration of saxagliptin and metformin IR tablets (Reference) formulations in fed state, linear mixed model analysis was performed on log[AUC(INF)] of metformin. Factors in the model were sequence, period and treatment as fixed effects, and participant within sequence as a random effect; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 6, analysis 2]; Mixed Models Analysis; Bioequivalence=90% CIs for the test; Geometric Mean Ratio, Test vs. Reference = 1.042, 90% CI 2-sided [0.986 to 1.102] — For AUC(INF) of metformin, the point estimate and 90% confidence interval (CI) were calculated for the ratio of the geometric mean of the Test formulation in fed state: the geometric mean of the Reference formulation in fed state

8. Primary Outcome: Metformin T-half and T-max
Description: T-half and T-max for single-dose metformin IR (500 mg), either coadministered with saxagliptin (2.5 mg), or administerd as FDC 2.5 mg saxagliptin/500 mg metformin IR, under fasted and fed conditions.
Time Frame: as for outcome 1
Population: PK data set, all participants who received study drug
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
hours
  T-Half | 9.87 (5.561) | 12.03 (9.014) | 8.62 (3.069) | 8.61 (3.288)
  T-max | 3.18 (0.919) | 3.08 (0.762) | 3.96 (0.204) | 3.87 (0.680)

9. Secondary Outcome: BMS-510849 Mean Cmax
Description: Cmax of the saxagliptin metabolite BMS-510849, following single-dose saxagliptin (2.5 mg) coadministered with metformin IR (500 mg) or administered as an FDC 2.5 mg saxagliptin/500 mg metformin IR tablet, under fasted and fed conditions.
Time Frame: as for outcome 1
Population: PK data set, all participants who received study drug
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng/mL | 16.32 (5.094) | 16.10 (4.967) | 18.40 (4.140) | 18.72 (4.280)

10. Secondary Outcome: BMS-510849 Mean AUC (0-T)
Description: AUC (0-T) for the saxagliptin metabolite BMS-510849, following single-dose saxagliptin (2.5 mg) coadministered with metformin IR (500 mg) or administration as an FDC 2.5 mg saxagliptin/500 mg metformin IR tablet, under fasted and fed conditions.
Time Frame: as for outcome 1
Population: PK data set, all participants who received study drug
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng*h/mL | 112.35 (20.053) | 113.87 (24.141) | 120.31 (22.719) | 123.05 (24.821)

11. Secondary Outcome: BMS-510849 Mean AUC (0-INF)
Description: AUC (0-T)= for the saxagliptin metabolite BMS-510849, following single-dose saxagliptin (2.5 mg) coadministered with metformin IR (500 mg) or administered as an FDC 2.5 mg saxagliptin/500 mg metformin IR tablet, under fasted and fed conditions.
Time Frame: as for outcome 1
Population: PK data set, all participants who received study drug
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng*h/mL | 120.72 (19.826) | 122.74 (24.805) | 129.02 (22.988) | 131.88 (25.908)

12. Secondary Outcome: BMS-510849 Mean T-half and T-max
Description: T-half and Tmax of the saxagliptin metabolite BMS-510849, following single-dose saxagliptin (2.5 mg) coadministered with metformin IR (500 mg) or administerd as an FDC 2.5 mg saxagliptin/500 mg metformin IR tablet, under fasted and fed conditions.
Time Frame: as for outcome 1
Population: PK data set, all participants who received study drug
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
hours
  T-Half | 6.53 (1.346) | 6.93 (1.284) | 6.73 (1.380) | 6.62 (1.238)
  T-max | 2.40 (0.965) | 2.30 (0.965) | 2.35 (0.774) | 2.53 (0.727)

13. Secondary Outcome: Number of Participants With at Least 1 Adverse Event (AE), Death, Serious AE (SAE), or AEs Leading to Discontinuation
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event.
Time Frame: From Day 1 through Day 45, including up to 56 days after last dose of study medication
Population: All Treated Participants
Measure: Number; unit: participants
Groups:
- Co-administration of Saxagliptin and Metformin IR (Fasted): Participants received oral co-administration of a 2.5 mg tablet of saxagliptin and a 500 mg tablet of metformin immediate release (IR) under fasted conditions
- Saxagliptin/Metformin (Fasted): Participants received a single oral dose of a fixed dose combination (FDC) tablet of 2.5 mg saxagliptin/500 mg metformin IR under fasting conditions
- Co-administration of Saxagliptin and Metformin IR (Fed): Participants received oral co-administration of a 2.5 mg tablet of saxagliptin and a 500 mg tablet of metformin immediate release (IR) under fed conditions
- Saxagliptin/Metformin (Fed): Participants received a single oral dose of a fixed dose combination (FDC) tablet of 2.5 mg saxagliptin/500 mg metformin IR under fed conditions
Arm/Group | Co-administration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin (Fasted) | Co-administration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin (Fed) | All Treated Participants
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
participants
  Participants with at least 1 AE | 6 | 3 | 4 | 1 | 7
  Death | 0 | 0 | 0 | 0 | 0
  SAE | 0 | 0 | 0 | 0 | 0
  AE leading to discontinuation | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Laboratory Marked Abnormalities
Description: High=greater than Upper Normal Limit (ULN), Low=lower than Lower Normal Limit (LLN). LLN/ULN= Leukocytes: <0.9 x LLN/ >1.2 x ULN; blood urea nitrogen (BUN): >1.1 x ULN; creatinine: >1.33 x BL; phosphorous (P): <0.75 x LLN/ >1.2 5 x ULN; creatinine kinase (CK): >1.5 x ULN; urine blood=use ≥2 x BL if value ≥2+ or BL1+
Time Frame: From Day 1 through Day 45, including up to 56 days after last dose of study medication
Population: All Treated Participants
Measure: Number; unit: participants
Arm/Group | Co-administration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin (Fasted) | Co-administration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin (Fed) | All Treated Participants
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
participants
  High leukocytes | 0 | 0 | 1 | 0 | 1
  High BUN | 0 | 1 | 0 | 0 | 1
  High creatinine | 0 | 0 | 1 | 0 | 1
  Low phosphorus | 0 | 1 | 0 | 0 | 1
  High CK | 0 | 0 | 1 | 0 | 1
  High urine blood | 0 | 1 | 0 | 0 | 1

15. Secondary Outcome: Number of Participants With Clinically Relevant Electrocardiogram (ECG) Abnormalities
Description: PR interval, QRS complex, width of QRS, QT interval, and QT corrected for heart rate adjusting for heart rate using either Bazett formula or Fridericia formula were measured. ECG abnormalities were judged to be of medical importance by the Investigator.
Time Frame: Period 1 Day 1, Period 2 Day 1, Period 3 Day 1, Period 4 Day 1, Period 4 Day 3
Population: All Treated Participants
Measure: Number; unit: participants
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
participants | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Clinically Relevant Vital Sign Abnormalities
Description: Mean systolic and diastolic blood pressure, heart rate, respiration, and temperature were assessed.Vital sign abnormalities abnormalities were judged to be of medical importance by the Investigator.
Time Frame: Period 1 Day 1, Period 2 Day 1, Period 3 Day 1, Period 4 Day 1, Period 4 Day 3
Population: All Treated Participants
Measure: Number; unit: participants
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
participants | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participant With Clinically Relevant Physical Examination Abnormalities
Description: A physical examination was conducted which included height and weight measurements, from which the Body Mass Index was determined. Physical examination abnormalities were judged to be of medical importance by the Investigator.
Time Frame: Screen, Period 1 Day -1, prior to discharge
Population: All Treated Participants
Measure: Number; unit: participants
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Number analyzed (Participants) | 24 | 24 | 24 | 24
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Saxagliptin/Metformin FDC (Fasted): Participants received a single oral dose of a fixed dose combination (FDC) tablet of 2.5 mg saxagliptin/500 mg metformin IR under fasting conditions
Arm/Group | Coadministration of Saxagliptin and Metformin IR (Fasted) | Saxagliptin/Metformin FDC (Fasted) | Coadministration of Saxagliptin and Metformin IR (Fed) | Saxagliptin/Metformin FDC (Fed)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 6/24 | 3/24 | 4/24 | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Coadministration of Saxagliptin and Metformin IR (Fasted) (N=24) | Saxagliptin/Metformin FDC (Fasted) (N=24) | Coadministration of Saxagliptin and Metformin IR (Fed) (N=24) | Saxagliptin/Metformin FDC (Fed) (N=24)
PALPITATIONS (Cardiac disorders) | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 1 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 0 | 0
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 0 | 0 | 0
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
INCREASED UPPER AIRWAY SECRETION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
FATIGUE (General disorders) | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.